CLINICAL TRIAL: NCT04735705
Title: A Prospective, Open-Label, Pilot, Multicentric Clinical Investigation to Evaluate the Performance and Safety of Cerviron Ovules® in the Local Treatment of Non-Specific or Endogenous, Symptomatic Vaginitis
Brief Title: Clinical Investigation To Evaluate Cerviron Ovules® in Symptomatic Vaginitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perfect Care Distribution (Industry)
Collaborators: MDX Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYRON/01/2021
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Vaginitis and Vulvovaginitis
Keywords: Vaginitis; vaginal discharge, vaginal pH, vaginal microflora
MeSH Terms: conditions — Vaginitis; Vulvovaginitis; Vaginal Discharge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerviron vaginal ovules (Experimental): Since Cerviron® has an innovative composition, we preferred an exploratory approach for the design of the present clinical investigation.
  Interventions: Device: Cerviron

INTERVENTIONS:
Device: Cerviron — Cerviron ovules ® is a class IIb medical device indicated as adjuvant in the treatment of acute and chronic vulvovaginitis of mechanical etiology, caused by changes of vaginal pH and changes of the vaginal flora. It is also used in cervical lesions of mechanical origin as it favors the healing and re-epithelialization processes and reduces the proliferation of endogenous pathogens.

SUMMARY:
CYRON is a Prospective, Open-Label, Pilot, Multicentric Clinical Investigation to Evaluate the Performance and Safety of Cerviron Ovules® in the Local Treatment of Non-Specific or Endogenous, Symptomatic Vaginitis. The primary objective is to assess the therapeutic performance and tolerability of Cerviron® Ovules in patients with symptomatic, non-specific, non-infectious vaginitis, and endogenous symptomatic infections.

The secondary objective of this clinical investigation is the assessment of performance of the medical device by several additionally clinical outcomes (vaginal discharge, vaginal pH, microscopic characteristics of inflammatory cells and characteristics of vaginal microflora).

Participants will also evaluate the degree of satisfaction related to the use of the medical device.

DETAILED DESCRIPTION:
Vaginitis is the general term characterizing a spectrum of disorders of the vagina caused by infection, inflammation, or changes in the normal vaginal flora. Symptoms include abnormal vaginal discharge, odour, pruritus, pain, dysuria and/or discomfort. Moreover, vaginitis is responsible for the most common problems in clinical medicine, and it is the reason cited most often for visits to obstetricians and gynecologists. In the past years, the problem of vaginitis has all too often been ignored by the medical community or regarded merely as a minor annoyance to women. According to Gardner, "Vaginitis must cause more unhappiness on earth than any other gynecologic disease. In addition to the many physical and emotional problems associated with vaginitis, the economic loss involved is of astronomic proportions." The most common causes of vaginitis are bacterial vaginosis, vulvovaginal candidiasis, and trichomoniasis. Bacterial Vaginosis is the cause in 40% to 50% of cases in which a cause is identified, with vulvovaginal candidiasis accounting for 20% to 25% and trichomoniasis for 15% to 20% of cases. The standard of care currently is based on anti-infectious therapy. With the availability of complementary and alternative therapies and over-the-counter medications for vaginitis, many symptomatic women seek these products before or in addition to an evaluation by a medical provider. However, recurrence of vaginosis is frequent, and can include four or more episodes in one year.

Non-infectious cases, including atrophic, irritant, and inflammatory vaginitis, are less common and account for 5% to 10% of vaginitis cases. Obtaining a medical history alone has been shown to be insufficient for accurate diagnosis of vaginitis and can lead to the inappropriate administration of medication. Therefore, a careful history, examination, and laboratory testing to determine the etiology of vaginal symptoms are needed. Information on sexual behaviors and practices, gender of sex partners, menses, vaginal hygiene practices (e.g., douching), and self-treatment with medications should be collected.

Other causes of vaginitis There is no cause of vagini¬tis identified in up to 30% of women. These women may have a range of conditions, includ¬ing irritant or allergic vaginitis, atrophic vaginitis, or physiologic discharge. The presence of objective signs of vulvar inflammation in the absence of vaginal pathogens after laboratory testing suggests the possibility of mechanical, chemical, allergic, or other non-infectious causes of vulvovaginal signs or symptoms.

Inflammatory vagi¬nitis is an uncommon condition characterized by purulent vaginal discharge, burning, and dyspa¬reunia, and should be considered in patients with these symptoms if no infectious cause is found. Inflammatory vaginitis is associated with low estrogen levels, such as in menopausal or perimenopausal women.

Desquamative inflammatory vaginitis is a chronic inflammatory process involving both vagina and vestibule, occurring almost exclusively in white women, that responds well to topical anti-inflammatory therapy. Long-term maintenance therapy is frequently required.

Irritant/allergic vaginitis is characterized by symptoms such as burning and soreness and signs such as vulvar erythema.

Atrophic vaginitis is an uncommon condition that occurs as a consequence of estrogen deficiency and is characterized by symptoms such as thin, clear discharge, vaginal dryness, dyspareunia, itching. An examination of the vulva can indicate inflammation and thin and friable vaginal mucosa. Risk factors contributing to atrophic vaginitis are menopause, lactation, oophorectomy, radiation therapy, chemotherapy, immunologic disorders, premature ovarian failure, endocrine disorders, and antioestrogen medications.

Aerobic vaginitis is a distinct vaginal condition, requiring different clinical management and with distinct clinical risks. (7) Aerobic vaginitis is defined by disruption in Lactobacillus dominance but is accompanied by more extreme inflammatory changes than BV and the presence of mainly aerobic enteric commensals or pathogens, including Group B Streptococcus (S. agalactiae), Enterococcus faecalis, Escherichia coli, and S. aureus. Streptococcus agalactiae (group B Streptococcus, GBS) vaginal pathogenicity is not uniformly acknowledged throughout the literature. GBS virulence for vagina was recognized in the past, as the organism has been observed to potentially cause local inflammation and discharge, as well as lactobacilli rarefaction.

Cytolitytic vaginosis is another condition which has been recently described as an entity distinct from either normal flora or bacterial vaginosis. This condition, also called Doderlein's vaginitis, has numerous, active lactobacilli damaging epithelial cells because of extreme acidity and low pH. The bare nuclei and cellular debris that are seen during microscopy, should not be mistaken for leucocytes and cocci.

Cerviron ovules® is a class IIb medical device indicated as adjuvant in the treatment of acute and chronic vulvovaginitis of mechanical etiology, caused by changes of vaginal pH and changes of the vaginal flora. It is also used in cervical lesions of mechanical origin as it favors the healing and re-epithelialization processes and reduces the proliferation of endogenous pathogens.

This is the first clinical investigation on human subjects with this medical device, in which 50 patients will be enlisted, and which will take place in two research centres in Romania.

ELIGIBILITY:
Inclusion Criteria:

* Adult females, aged 18 years to 65 years;
* Subjects presenting two or more vaginal symptoms such as leucorrhoea, pruritus, burning sensation, erythema, pain, odour, dysuria, or dyspareunia;
* Subjects with a diagnosis of either non-infectious vaginitis, or endogenous, symptomatic infection;
* Negative for Gardnerella vaginalis, Candida albicans, Trichomonas vaginalis;
* Subjects willing to provide signed informed consent to clinical investigation participation.

Exclusion Criteria:

* Subjects in menstrual period or suffering from menorrhagia;
* Colpectomy;
* Subjects with undiagnosed abnormal genital bleeding;
* Subject with vulvar, vaginal or cervical cancer;
* Known, active sexually transmitted infection (STI) in partner, as per anamnesis;
* Subjects with HIV or other immunodeficiency;
* Subjects with any pathology of the female reproductive organs;
* Known allergy or hypersensitivity to the medical device ingredients;
* Use of spermicides;
* Use of diaphragm;
* Concomitant topical or systemic anti-infective treatment;
* Unable to comply with visit procedures;
* Subjects included in other clinical investigations;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramona Petrita, CSO, Study Director — MDX Research
Locations (2):
- Romania (2):
  - Spitalul Clinic Județean de Urgență "Pius Brinzeu", Timișoara, Timiș County
  - Institutul National pentru Sanatatea Mamei si Copilului (INSMC) "Alessandrescu - Rusescu", Bucharest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toader DO, Olaru RA, Iliescu DG, Petrita R, Calancea FL, Petre I. Clinical Performance and Safety of Vaginal Ovules in the Local Treatment of Nonspecific Vaginitis: A National, Multicentric Clinical Investigation. Clin Ther. 2023 Sep;45(9):873-880. doi: 10.1016/j.clinthera.2023.06.023. Epub 2023 Jul 18. PMID 37474354

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cerviron Vaginal Ovules
Started | 50
Completed | 47
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cerviron Vaginal Ovules
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.23 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Childbirth potential [Count of Participants; unit: Participants] | 36
Subject in menopause [Count of Participants; unit: Participants] | 9
Subject pregnant [Count of Participants; unit: Participants] | 0
History of cancer [Count of Participants; unit: Participants] | 2
Sex life [Count of Participants; unit: Participants] — Active sex life
  Participants | 44
Reproductive life [Count of Participants; unit: Participants] | 25
Tobacco consumption [Count of Participants; unit: Participants] | 20
Alcohol consumption [Count of Participants; unit: Participants] | 0
Physical activity [Count of Participants; unit: Participants] | 32
Rest/Day [Count of Participants; unit: Participants] — Rest/day (7-8 hours)
  Participants | 34
Hydration [Count of Participants; unit: Participants] — Hydration/day (1,5-2 L of water)
  Participants | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Same Gynaecological Conditions at the End of Treatment Visit
Description: Success is defined by resolution (return to patient's usual gynaecological conditions, i.e. before the episode which warranted inclusion in the study) OR substantial improvement of clinical signs of infectious vaginitis (i.e. abnormal vaginal discharge), and/or vaginal symptoms (vaginal burning and/or vaginal pain, and/or vaginal irritation and/or pruritus and/or odor). Failure is defined by persistence or worsening of symptoms and clinical signs or requirement of an alternative or specific treatment.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cerviron Vaginal Ovules
Number analyzed (Participants) | 47
Participants | 13

2. Primary Outcome: Rate of Treatment-related Adverse Events in Subjects Participating in the Clinical Investigation
Description: The safety of CERVIRON ® as measured by the rate of treatmentrelated adverse events, including serious adverse events (SAEs), in subjects participating in the clinical investigation.
Time Frame: 3 months
Measure: Number; unit: AEs
Arm/Group | Cerviron Vaginal Ovules
Number analyzed (Participants) | 47
AEs | 3

3. Secondary Outcome: Number of Participants With Absent, Mild, Moderate or Abundant Vaginal Discharge at 1, 2 and 3 Months of Treatment
Description: The vaginal discharge assessed by the investigator by using a score:
  0=absent
  1. mild: insufficient for speculum collection
  2. moderate: sufficient for speculum collection
  3. abundant: visible at the introitus even before speculum introduction
  4. purulent, abnormal discharge: visible at the introitus even before speculum introduction
Time Frame: at 1, 2 and 3 months
Measure: Number; unit: participants
Arm/Group | Cerviron Vaginal Ovules
Number analyzed (Participants) | 47
participants
  Absent - 1 month | 2
  Absent - 2 months | 8
  Absent - 3 months | 9
  Mild - 1 month | 26
  Mild - 2 months | 21
  Mild - 3 months | 13
  Moderate - 1 month | 19
  Moderate - 2 months | 18
  Moderate - 3 months | 25
  Abundant - 1 month | 0
  Abundant - 2 months | 0
  Abundant - 3 months | 0
  Purulent - 1 month | 0
  Purulent - 2 months | 0
  Purulent - 3 months | 0

4. Secondary Outcome: Number of Participants With Change in Vaginal pH Values
Description: Determination of pH values compared to its normal values (3.8 - 4.5)
Time Frame: at 1, 2 and 3 months
Measure: Number; unit: Participants
Arm/Group | Cerviron Vaginal Ovules
Number analyzed (Participants) | 47
Participants
  Normal - 1 month | 41
  Normal - 2 months | 44
  Normal - 3 months | 47
  Abnormal - 1 month | 6
  Abnormal - 2 months | 3
  Abnormal - 3 months | 0

5. Secondary Outcome: Number of Participants With Change in Vaginal Microflora and Lactobacilli Count
Description: The change in Lactobacillus species as shown by microscopy
Time Frame: 3 months
Measure: Number; unit: Participants
Arm/Group | Cerviron Vaginal Ovules
Number analyzed (Participants) | 47
Participants
  Lactobacilli present | 30
  Leukocytes present | 38
  Enterobact. present | 0
  Squamous epithelial cells present | 0
  Gardnerella vaginalis present | 2
  Trich. vaginalis present | 0
  Candida present | 2
  Yeast cells and filaments present | 2

6. Secondary Outcome: Number of Participants With Change in Vaginal Inflammation
Description: The change in inflammatory and parabasal cells by microscopy
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cerviron Vaginal Ovules
Number analyzed (Participants) | 47
Participants | 32

7. Secondary Outcome: Results in Patient Satisfaction's Scale (Likert Scale)
Description: The degree of satisfaction when using the medical device will be assessed using a five-point Likert Scale. The degree of satisfaction when using the medical device was assessed using a five-point Likert Scale, as very satisfied, satisfied, neutral, unsatisfied, and very unsatisfied.
Time Frame: 3 months
Measure: Number; unit: Participants
Arm/Group | Cerviron Vaginal Ovules
Number analyzed (Participants) | 47
Participants
  Very Satisfied | 39
  Satisfied | 6
  Neutral | 2
  Unsatisfied | 0
  Very Unsatisfied | 0

ADVERSE EVENTS:
Time Frame: During all the clinical investigation
Description: No significant adverse events (AEs) were reported during this clinical investigation.
Arm/Group | Cerviron Vaginal Ovules
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 3/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cerviron Vaginal Ovules (N=47)
Streptococcus infection (Infections and infestations) | 1 (1)
E. Coli infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT04735705/Prot_SAP_000.pdf